CLINICAL TRIAL: NCT03589976
Title: A Single Center Randomized,Double Blind, Placebo-controlled Futility Trial to Determine if Sirolimus is of Sufficient Promise to Slow the Progression of Multiple System Atrophy
Brief Title: A Futility Trial of Sirolimus in Multiple System Atrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis showed early evidence of futility of sirolimus. Trial stopped per DSMB recommendation.
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 17-01392
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus (Experimental): 2 mg/day (one 2-mg tablet/day). The dose of sirolimus will be adjusted throughout the trial based on sirolimus plasma levels and the presence of drug-related adverse events. The maximum dose of sirolimus will be6 mg/day (three 2-mg tablets/day).
  Interventions: Drug: Sirolimus 2 MG
- Placebo (Placebo Comparator): Patients receiving placebo will undergo analog sham level measurements and the number of tablets will be also adjusted to maintain the blinding of the trial.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sirolimus 2 MG — Dose will be adjusted throughout this trial based on sirolimus plasma levels and the presence of drug-related adverse events. The maximum dose will be 6mg/day.
  Arms: Sirolimus
Other: Placebo — Patients receiving placebo will undergo analog sham level measurements and the number of tablets will be also adjusted to maintain the blinding of the trial.
  Arms: Placebo

SUMMARY:
Single-center, randomized, placebo-controlled, phase-II, futility clinical trial to determine if oral sirolimus is of sufficient promise to slow disease progression in MSA, prior to embarking on a large-scale and costly phase III study to assess its efficacy. A futility design under the null hypothesis assumes that sirolimus will slow the progression of the disease, whereas the alternative hypothesis assumes no benefit of sirolimus. If the null hypothesis is rejected (i.e., futility of sirolimus to slow progression of MSA), a major phase III study will be discouraged, whereas non-futility will offer strong support for a phase III trial to detect clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 30-80 years old with a diagnosis of MSA based on clinical criteria and standardized autonomic testing. This approach allows for identification of patients with MSA with very high specificity and is yet sensitive enough to allow for enrollment of patients at a disease stage at which an intervention on the natural disease course has a meaningful impact on patient outcome. Patients therefore have to fulfill current consensus criteria (1) for probable MSA of the parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C) and have findings on autonomic function testing suggestive of MSA.
* Participants who are less than 4 years from the time of documented MSA diagnosis.
* Participants who are still able to walk with or without assistance.
* Participants with an anticipated survival of at least 3 years in the opinion of the investigator.
* Participants who are willing and able to give informed consent.
* Montreal Cognitive Assessment (MoCA) > 20.
* Ability to take oral medication and be willing to adhere to the study drug regimen
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 8 weeks after the end of study drug administration
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

* Women of childbearing potential who do not practice an acceptable method of birth control. Acceptable methods of birth control in this study are: surgical sterilization, intrauterine devices, partner's vasectomy, a double-protection method (condom or diaphragm with spermicide), hormonal contraceptive drug (i.e., oral contraceptive, contraceptive patch, long-acting injectable contraceptive) with a required second mode of contraception.
* Participants with a clinically significant or unstable medical or surgical condition that, in the opinion of the investigator, might preclude safe completion of the study or might affect the results of the study. These include conditions causing significant central nervous system (CNS) or autonomic dysfunction, including congestive heart failure, recent (<6 months) myocardial infarct, cardiopulmonary disease, severe, uncontrolled hypertension, thrombocytopenia (< 50 x 10(9)/L), severe anemia (< 8g/dl), immunocompromised state, liver or kidney disease (creatinine > 1.5 mg/dl or proteinuria > 20 mg/dl), uncontrolled diabetes mellitus (HbA1c >10g%), alcoholism, amyloidosis, uncontrolled hypothyroidism, sympathectomy, unstable peripheral neuropathies, concurrent infections, orthopedic problems that compromise mobility and activity of daily living, cerebrovascular accidents, neurotoxin or neuroactive drug exposure, parkinsonism due to drugs (including neuroleptics, alpha-methyldopa, reserpine, metoclopramide).
* Participants with high LDL cholesterol levels (LDL > 160 mg/dL) and/or high triglycerides levels (> 200 mg/dL).
* Participants with latent tuberculosis infection as defined as positive interferon-gamma release-assay (QUANTIferon®).
* Participants with history of tuberculosis
* Participants with a history of active, acute or chronic, or latent hepatitis B or hepatitis C.
* Participants with human immunodeficiency virus (HIV) infection, or other congenital or acquired causes of immunosuppression.
* Participants with active malignant neoplasms or history of malignant neoplasm in the last 5 years.
* Movement disorders other than MSA; e.g., Parkinson disease, dementia with Lewy bodies, essential tremor, progressive supranuclear palsy, spinocerebellar ataxia, spastic paraparesis, corticobasal degeneration, or vascular, pharmacological or post-encephalitic parkinsonism.
* Dementia (DSM-V criteria).
* History of electroconvulsive therapy.
* History of deep brain stimulation surgery.
* Patients with contraindication for MRI scanning, including those with MRI-incompatible pacemaker
* History of organ transplant
* Participants who have taken any investigational products within 60 days prior to baseline.
* Treatment with cyclosporine, corticosteroids, methotrexate, rituximab within 3 months prior to baseline.
* Treatment with inhibitors of CYP3A4 (which may decrease the metabolism of sirolimus and increase sirolimus levels): nicardipine, verapamil, clotrimazole, fluconazole, itraconazole, clarithromycin, erythromycin, troleandomycin, cisapride, metoclopramide, bromocriptine, cimetidine, danazol, HIV-protease inhibitors (e.g., ritonavir, indinavir); grapefruit.
* Treatment with inducers of CYP3A4 (which may increase the metabolism of sirolimus and decrease sirolimus levels): carbamazepine, phenobarbital, phenytoin, rifabutin, rifapentine.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Alberto Palma, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal that has been approved by a local Institutional Review Board.

REFERENCES:
- [Derived] Palma JA, Martinez J, Millar Vernetti P, Ma T, Perez MA, Zhong J, Qian Y, Dutta S, Maina KN, Siddique I, Bitan G, Ades-Aron B, Shepherd TM, Kang UJ, Kaufmann H. mTOR Inhibition with Sirolimus in Multiple System Atrophy: A Randomized, Double-Blind, Placebo-Controlled Futility Trial and 1-Year Biomarker Longitudinal Analysis. Mov Disord. 2022 Apr;37(4):778-789. doi: 10.1002/mds.28923. Epub 2022 Jan 18. PMID 35040506

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus | Placebo
Started | 35 | 12
Completed | 16 | 6
Not Completed | 19 | 6
Not completed — Death | 5 | 1
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus | Placebo | Total
Number analyzed (Participants) | 35 | 12 | 47
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [56 to 63] | 58 [56 to 63] | 58 [56 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 21 | 6 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 33 | 11 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 30 | 12 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 12 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 48 Weeks in United Multiple System Atrophy Rating Score (UMSARS) Total Score
Description: UMSARS is a validated, disease-specific scale representing the diverse signs and symptoms in MSA.
  USMARS has an Activities of Daily Living score (UMSARS-1, 12 questions) that evaluates motor including autonomic activities and the Motor Examination score (UMSARS-2, 14 questions). UMSARS-3 measures supine/standing BP and UMSARS-4 is a disability scale.
  The total range of score is 1-109; Higher scores on the UMSARS scales mean poorer health.
Time Frame: Baseline, 48 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 25 | 9
score on a scale | 13.92 (8.32) | 11.3 (8)

2. Secondary Outcome: Change From Baseline to 48 Weeks in UMSARS-1
Description: The Activities of Daily Living score (UMSARS-1, 12 questions) evaluates impact of symptoms, including autonomic, on activities of daily living.
  12 functional situations are rated between 0-4. The total range of score is 0-48; the higher the score, the more problems conducting activities of daily living.
Time Frame: Baseline, 48 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 25 | 9
score on a scale | 5.65 (5.91) | 5.33 (3.81)

ADVERSE EVENTS:
Time Frame: month 12 after initiation of study drug) (+ 15 days)
Arm/Group | Sirolimus | Placebo
All-Cause Mortality (participants affected / at risk) | 5/35 | 1/12
Serious Adverse Events (participants affected / at risk) | 9/35 | 2/12
Other Adverse Events (participants affected / at risk) | 31/35 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=35) | Placebo (N=12)
Death (General disorders) | 5 | 1
Other (General disorders) | 4 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=35) | Placebo (N=12)
Infections (Infections and infestations) | 21 | 4 — Urinary tract infection, upper respiratory infection, skin infection, sinus infection
Aphthae, gingivitis, and oral herpes-like vesicles (Skin and subcutaneous tissue disorders) | 15 | 2
Diarrhea (Gastrointestinal disorders) | 16 | 2
Edema in Lower Limbs (Vascular disorders) | 17 | 1
Acne, Petechiae, Rash (Skin and subcutaneous tissue disorders) | 13 | 2
Fall (Nervous system disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 3 | 1
Worsening of Movement Disorder (Nervous system disorders) | 4 | 1
Fatigue (General disorders) | 1 | 7
Other (General disorders) | 25 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT03589976/Prot_SAP_000.pdf